CLINICAL TRIAL: NCT05940649
Title: Continuous Versus Bolus Administration of Norepinephrine to Treat Hypotension During Anesthetic Induction - the INDUCT Randomized Trial
Brief Title: Continuous Versus Bolus Administration of Norepinephrine to Treat Hypotension During Anesthetic Induction
Acronym: INDUCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kristen Thomsen (Other)
Responsible Party: Sponsor-Investigator, Kristen Thomsen, Dr., Universitätsklinikum Hamburg-Eppendorf
Organization: Universitätsklinikum Hamburg-Eppendorf (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2023-100999-BO-ff
Record Dates: First submitted 2023-07-04; First posted 2023-07-11 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Intraoperative Hypotension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuous norepinephrine administration (Experimental)
  Interventions: Procedure: Continuous norepinephrine administration
- Bolus norepinephrine administration (No Intervention)

INTERVENTIONS:
Procedure: Continuous norepinephrine administration — In patients randomized to continuous norepinephrine administration, hypotension (= mean arterial pressure < 65mmHg) will be treated with continuous norepinephrine infusion. The norepinephrine perfusion line will be connected to the saline infusion line using a three-way valve. Treating anesthesiologists will be free to reduce or increase the norepinephrine infusion rate anytime.
  Arms: Continuous norepinephrine administration

SUMMARY:
Intraoperative hypotension is common in patients having non-cardiac surgery with general anesthesia and is associated with organ injury and death. The timely treatment of intraoperative hypotension is thus important to avoid postoperative complications. About one third of intraoperative hypotension occurs during anesthetic induction - i.e., between the start of anesthetic induction and surgical incision. Hypotension during anesthetic induction is associated with postoperative acute kidney injury.

Unmodifiable risk factors for hypotension during anesthetic induction include age, male sex, and a high American Society of Anesthesiologists physical status class. However, hypotension during anesthetic induction is mainly driven by modifiable factors - specifically, anesthetic drugs that cause vasodilation.

In most German hospitals, norepinephrine is the first-line vasopressor to treat hypotension during anesthetic induction. Norepinephrine is usually given as repeated manual boluses of 5, 10, or 20 μg. The continuous administration of norepinephrine via a perfusion pump is usually started only later. It remains unknown whether giving norepinephrine continuously - compared to giving it as repeated manual boluses - reduces hypotension during anesthetic induction.

We thus propose to investigate whether giving norepinephrine continuously - compared to giving it as repeated manual boluses - reduces hypotension during anesthetic induction in non-cardiac surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* non-cardiac surgery
* >45 years of age
* American Society of Anesthesiologists physical status classification II, III, and IV.

Exclusion Criteria:

* Planned intraarterial blood pressure monitoring during anesthetic induction with an arterial catheter
* Emergency surgery
* Transplant surgery
* History of organ transplant
* Pregnancy
* Heart rhythms other than sinus rhythm
* Impossible Finger-cuff blood pressure monitoring
* Rapid sequence induction

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Hypotension during anesthetic induction | First 15 minutes of anesthetic induction
  Area under a MAP of 65 mmHg [mmHg x min]

SECONDARY OUTCOMES:
Hypotension during anesthetic induction | First 15 minutes of anesthetic induction
  Area under a MAP of 60, 50, and 40 mmHg [mmHg x min]
Hypotension during anesthetic induction | First 15 minutes of anesthetic induction
  Duration of a MAP <65, <60, <50, and <40 mmHg [min]
Hypertension during anesthetic induction | First 15 minutes of anesthetic induction
  Duration of a MAP >100, >110, >120, and >140 mmHg [min]
Hypertension during anesthetic induction | First 15 minutes of anesthetic induction
  Area above a MAP of 100, 110, 120, and 140 mmHg [mmHg x min]
Hypertension during anesthetic induction | First 15 minutes of anesthetic induction
  Absolute [n] and relative [%] number of patients with any MAP measurement >100, >110, >120 and >140 mmHg
Hypotension during anesthetic induction | First 15 minutes of anesthetic induction
  Absolute [n] and relative [%] number of patients with any MAP measurement <65, <60, <50, and <40 mmHg
Hypotension during anesthetic induction | First 15 minutes of anesthetic induction
  Absolute [n] and relative [%] number of patients with at least one 1-minute episode of a MAP <65, <60, <50, and <40 mmHg
Hypotension during anesthetic induction | First 15 minutes of anesthetic induction
  Cumulative dose of norepinephrine indexed to body weight [μg kg-1]

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No